CLINICAL TRIAL: NCT01274130
Title: Investigatory Study of Metformin's Pharmacokinetics, Pharmacodynamics and Drug Drug Interactions Classifying the Group by MATE1 Genotype in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 4-2010-0417
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Adult
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranitidine (Experimental)
  Interventions: Drug: Metformin
- Verapamil (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Diavex 1000mg on Day1 and 750mg on Day2
  Other Names: Diavex®

SUMMARY:
This is the investigatory study to find out metformin's pharmacokinetics, pharmacodynamics and drug-drug interactions classifying the group by MATE1 genotype in healthy volunteers. The investigators will apply ranitidine and verapamil to the drug interaction study of metformin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 20 to 50 years at screening
* Subjects whose weights are heavier than or equal to 50 kg and ±20% of ideal body weight : Ideal body weight = (height cm - 100) x 0.9
* Subjects who provided written, voluntary informed consent to participate in this clinical trial and to comply the directions including contraception after being fully informed of and understand this trial

Exclusion Criteria:

* Subjects who have the clinically significant diseases or history in liver, kidney, nervous system, respiratory system, endocrine system, blood tumor and cardiovascular system.
* Subjects who have participated in other clinical trial within 1 month prior to the first day of drug administration
* Subjects who are inappropriate in the judgement of the investigator due to the reasons including clinical laboratory test results

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea